CLINICAL TRIAL: NCT06057896
Title: Combined Natural Molecules Improve Markers of Metabolic Syndrome and Climacteric in Menopausal Women
Brief Title: Effects of Combined Natural Molecules on Metabolic Syndrome in Menopausal Women
Status: Completed | Type: Observational
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Other Study IDs: Ins-SM-23
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-09

CONDITIONS: Menopause; Climacteric Syndrome; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Inositol; Phytoestrogens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- inositol, phytoestrogens, cocoa polyphenols
  Interventions: Dietary Supplement: inositol, phytoestrogens, cocoa polyphenols

INTERVENTIONS:
Dietary Supplement: inositol, phytoestrogens, cocoa polyphenols — myo-inositol, soy isoflavones and cocoa polyphenols

SUMMARY:
The study collected retrospective data from the assumption of combined natural molecules in menopausal women with metabolic syndrome

ELIGIBILITY:
Inclusion Criteria:

* menopause
* diagnosis of metabolic syndrome

Exclusion Criteria:

* pharmacologically-induced menopause
* hormonal therapies
* sensitizing insulin therapies
* cancer patient or ex-cancer patient

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women in menopause exhibiting at least three of the diagnostic criteria for metabolic syndrome
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Body mass index | [0, 6 months]
  Change of body weight

SECONDARY OUTCOMES:
Climacteric | [0, 6 months]
  Changes of number of flushes
Climateric | [0, 6 months]
  Changes of intensity of flushes measured through questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mario Passaro, MD, Principal Investigator — ASL NA3 Sud, Naples, Italy.
Locations (1):
- SCCAL, Naples, Italy